CLINICAL TRIAL: NCT00330447
Title: Oncological Treatment During Pregnancy: Pharmacokinetics of Chemotherapy and Long Term Follow up of the Offspring
Brief Title: Effects of Oncological Treatment During Pregnancy on Mother and Child
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: The Netherlands Cancer Institute (Other); Erasmus Medical Center (Other); San Gerardo Hospital (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Frederic Amant, MD, PhD, University Hospital, Gasthuisberg
Other Study IDs: cancer in pregnancy
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cancer; Pregnancy
Keywords: pregnancy; in utero; chemotherapy; radiotherapy; cancer; offspring; neonatal; long term; follow up; cancer during pregnancy; chemotherapy and radiotherapy during pregnancy; long term follow up of children
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Biospecimen Retention: Samples With DNA — Maternal blood serum and sediment of blood; from 2010 on we collect umbilical cord blood.
  Since new approval of protocol version 4.2 (08-02-2018) we collect samples of placental tissue, umbilical cord tissue and membranes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Studygroup: Cancer in Pregnancy - all diagnoses and treatments Children born from mothers diagnosed with cancer during pregnancy
- Control group: Children from the general population

SUMMARY:
The researchers aim to investigate the outcome (overall survival) of mothers who are diagnosed and/or treated for cancer during pregnancy. Furthermore they want to test the hypothesis that children who were exposed to cancer or cancer treatment (cytotoxic drugs, radiation therapy, targeted therapy,...) develop normally (neurologic and cardiologic examination).

DETAILED DESCRIPTION:
Study contains several study parts (protocol version 4.4):

**********Part I. Pregnancy, delivery and maternal health********** Part I.I.A. Registration study 'Cancer during pregnancy' mother and neonate None Part I.I.B. Effects of prenatal exposure to cancer treatment on fetal growth. The association between placental pathophysiologic mechanisms (histopathology and immunohistochemistry), circulating maternal factors and fetal growth.

From participating women, a maternal blood sample will be collected during or shortly after birth. Also, an umbilical cord blood sample and placental and umbilical cord biopsies will be drawn.

Part I.II. Measurement of maternal and paternal anxiety and emotional needs when confronted with a cancer diagnosis during pregnancy The participants will be asked to complete questionnaires.

**********Part II. Child********** Long term follow up of children and adolescents in utero exposed to chemotherapy and/or radiotherapy Regular check-ups of the child, at the age of 6 months, 18 months, 3y, 6y, 9y, 12y, 15y, and 18y, and after the age of 18 years: 5-yearly cardiologic assessment and questionnaires (23y, 28y, 33y, 38y, and 43y). Optional at the ages of 9y, 12y, 15y and 18y: MRI session.

Summary part I:

Prospectively the outcome of mothers diagnosed and/or treated for cancer during pregnancy will be registered and investigated.

Summary Part II:

In a prospective trial we invite children that were exposed to cytotoxic drugs or radiotherapy in utero for a standardized neurological and cardiological examination. The examinations will be done by qualified psychologists, neurological and cardiological pediatricians.

ELIGIBILITY:
Patients do not need to participate in both; however, preferentially both study parts should be performed.

**************Part I: Pregnancy, delivery and maternal health**************

Patients must meet the following inclusion criteria:

* Histologically proven cancer in association with a pregnancy (during pregnancy or cancer dagnosis within 5 years after pregnancy)
* > 18 years of age, premenopausal
* Patients who have given their signed and written informed consent to participate in the trial after fully understanding the implication of the protocol
* Women receiving any cytotoxic drug or radiation therapy during pregnancy are allowed for the assessment of the maternal and fetal outcome (Part II).

Exclusion Criteria:

* Mentally disabled or significantly altered mental status that would prohibit the understanding and giving of informed consent

**************Part II: Follow-up of children**************

Inclusion Criteria:

- Children that were prenatally exposed to cancer of cancer treament. Informed Consent is asked from parents. From the age of 12 years, informed assent is additionally asked from the child. After the age of 18 years, informed consent is solely asked of the offspring.

Exclusion Criteria:

* Mentally disabled or significantly altered mental status that would prohibit the understanding and giving of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Premenopausal women with a cancer diagnosis in association with cancer
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2005-08 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Follow-up of the mothers diagnosed with cancer during pregnancy | anticipated
  treatment during pregnancy, obstetrical outcome, maternal survival
Follow-up of the children antenatally exposed to chemotherapy or radiotherapy | anticipated
  neurologic and cardiologic outcome

CONTACTS AND LOCATIONS:
Overall Officials: Amant Frederic, MD PhD, Principal Investigator — KULeuven, Belgium
Locations (33):
- Cooper University Hospital (2015-ongoing), Camden, New Jersey, United States
- Instituto Alexander Fleming, Buenos Aires, Argentina
- Universitätsklinik für Frauenheilkunde und Geburtshilfe (retrospective 2016-2018), Graz, Austria
- Belgium (2):
  - UCL Brussels (2013-ongoing), Brussels
  - UZ Gasthuisberg, Katholieke Universiteit Leuven (2004-ongoing), Leuven
- Czechia (2):
  - University Hospital Ostrava (2018-ongoing), Ostrava
  - 3rd medical faculty of Charles University (2010-ongoing), Prague
- Copenhagen University Hospital (2015-ongoing), Copenhagen, Denmark
- Hopital Bichat-Claude-Bernard (retrospective until 2018), Paris, France
- Universitätsklinik Freiburg (retrospective until 2018), Freiburg im Breisgau, Germany
- Greece (4):
  - Euroclinic Hospital (2016-ongoing), Athens
  - Hellenic Anticancer-Oncological Hospital of Athens (retrospective 2015-2018), Athens
  - Ioannina University Hospital (retrosepctive 2015-2018), Ioannina
  - Hippokration Hospital (retrospective 2015-2018), Thessaloniki
- Italy (5):
  - European Institute of Oncology (2010-ongoing), Milan
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore (2012-ongoing), Milan
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico Milano (2017-ongoing), Milan
  - San Raffaele Hospital (2017-ongoing), Milan
  - CIttà della Salute e della Scienza di Torino (2015-ongoing), Torino
- Regional Hospital of High Specialty of Ixtapaluca (2018-ongoing), Ixtapaluca, Mexico
- Erasmus Medical Center (2014-ongoing), Rotterdam, Netherlands
- Haukeland University Hospital (2017-ongoing), Bergen, Norway
- Poland (3):
  - Medyczne Macierzynstwo (retrospective 2010-2018), Krakow
  - University Hospital Krakow (2018-ongoing), Krakow
  - Pozanan University of Medical Sciences (2017-ongoing), Poznan
- Hospital de Vila Franca de Xira (2017-ongoing), Vila Franca de Xira, Portugal
- Russia (3):
  - N.N.Blokchin National Medical Research Center of Oncology (2013-2018 retrospective; 2018-ongoing prospective), Moscow
  - Research Center for Obstetrics, Gynecology and Perinatology (2014-ongoing), Moscow
  - Almazov National Medical Research Center (2018-ongoing), Saint Petersburg
- Karolinska University Hospital (2017-ongoing), Stockholm, Sweden
- F.Hached University Teaching Hospital (retrospective 2016-2018), Sousse, Tunisia
- Trakya University Faculty of Medicine (retrospective 2015-2018), Edirne, Turkey (Türkiye)
- Grigoriev Institute for medical Radiology (retrospective until 2018), Kharkiv, Ukraine

REFERENCES:
- [Background] Caluwaerts S, VAN Calsteren K, Mertens L, Lagae L, Moerman P, Hanssens M, Wuyts K, Vergote I, Amant F. Neoadjuvant chemotherapy followed by radical hysterectomy for invasive cervical cancer diagnosed during pregnancy: report of a case and review of the literature. Int J Gynecol Cancer. 2006 Mar-Apr;16(2):905-8. doi: 10.1111/j.1525-1438.2006.00223.x. PMID 16681782
- [Background] Van Calsteren K, Berteloot P, Hanssens M, Vergote I, Amant F, Ganame J, Claus P, Mertens L, Lagae L, Delforge M, Paridaens R, Noens L, Humblet Y, Vandermeersch B, De Muylder X. In utero exposure to chemotherapy: effect on cardiac and neurologic outcome. J Clin Oncol. 2006 Apr 20;24(12):e16-7. doi: 10.1200/JCO.2006.06.1382. No abstract available. PMID 16622256
- [Background] Lishner M, Avivi I, Apperley JF, Dierickx D, Evens AM, Fumagalli M, Nulman I, Oduncu FS, Peccatori FA, Robinson S, Van Calsteren K, Vandenbroucke T, Van den Heuvel F, Amant F. Hematologic Malignancies in Pregnancy: Management Guidelines From an International Consensus Meeting. J Clin Oncol. 2016 Feb 10;34(5):501-8. doi: 10.1200/JCO.2015.62.4445. Epub 2015 Nov 30. PMID 26628463
- [Background] Amant F, Verheecke M, Wlodarska I, Dehaspe L, Brady P, Brison N, Van Den Bogaert K, Dierickx D, Vandecaveye V, Tousseyn T, Moerman P, Vanderstichele A, Vergote I, Neven P, Berteloot P, Putseys K, Danneels L, Vandenberghe P, Legius E, Vermeesch JR. Presymptomatic Identification of Cancers in Pregnant Women During Noninvasive Prenatal Testing. JAMA Oncol. 2015 Sep;1(6):814-9. doi: 10.1001/jamaoncol.2015.1883. PMID 26355862
- [Background] de Haan J, Verheecke M, Amant F. Management of ovarian cysts and cancer in pregnancy. Facts Views Vis Obgyn. 2015;7(1):25-31. PMID 25897369
- [Background] Amant F, Han SN, Gziri MM, Vandenbroucke T, Verheecke M, Van Calsteren K. Management of cancer in pregnancy. Best Pract Res Clin Obstet Gynaecol. 2015 Jul;29(5):741-53. doi: 10.1016/j.bpobgyn.2015.02.006. Epub 2015 Mar 4. PMID 25797199
- [Background] van Dam L, Han SN, Dierickx D, Amant F. Optimal staging of lymphoma during pregnancy is crucial. Womens Health (Lond). 2015 Mar;11(2):101-2. doi: 10.2217/whe.14.77. No abstract available. PMID 25776282
- [Background] Han SN, Van Peer S, Peccatori F, Gziri MM, Amant F; International Network on Cancer, Infertility and Pregnancy. Contraception is as important as fertility preservation in young women with cancer. Lancet. 2015 Feb 7;385(9967):508. doi: 10.1016/S0140-6736(15)60201-X. No abstract available. PMID 25705843
- [Background] Han SN, Verheecke M, Vandenbroucke T, Gziri MM, Van Calsteren K, Amant F. Management of gynecological cancers during pregnancy. Curr Oncol Rep. 2014 Dec;16(12):415. doi: 10.1007/s11912-014-0415-z. PMID 25344340
- [Background] Van Calsteren K, Amant F. Cancer during pregnancy. Acta Obstet Gynecol Scand. 2014 May;93(5):443-6. doi: 10.1111/aogs.12380. PMID 24628416
- [Background] Amant F, Halaska MJ, Fumagalli M, Dahl Steffensen K, Lok C, Van Calsteren K, Han SN, Mir O, Fruscio R, Uzan C, Maxwell C, Dekrem J, Strauven G, Mhallem Gziri M, Kesic V, Berveiller P, van den Heuvel F, Ottevanger PB, Vergote I, Lishner M, Morice P, Nulman I; ESGO task force 'Cancer in Pregnancy'. Gynecologic cancers in pregnancy: guidelines of a second international consensus meeting. Int J Gynecol Cancer. 2014 Mar;24(3):394-403. doi: 10.1097/IGC.0000000000000062. PMID 24445819
- [Background] Vandenbriele C, Dierickx D, Amant F, Delforge M. The treatment of hematologic malignancies in pregnancy. Facts Views Vis Obgyn. 2010;2(2):74-87. No abstract available. PMID 25302102
- [Background] Deckers S, Amant F. Breast cancer in pregnancy: a literature review. Facts Views Vis Obgyn. 2009;1(2):130-41. PMID 25478078
- [Background] Gziri MM, Goffin F, Debieve F, Amant F. [Cancer diagnosis during pregnancy: importance of a national and European registration]. Rev Med Liege. 2013 Oct;68(10):527-30. French. PMID 24298727
- [Background] Han SN, Kesic VI, Van Calsteren K, Petkovic S, Amant F; ESGO 'Cancer in Pregnancy' Task Force. Cancer in pregnancy: a survey of current clinical practice. Eur J Obstet Gynecol Reprod Biol. 2013 Mar;167(1):18-23. doi: 10.1016/j.ejogrb.2012.10.026. Epub 2012 Nov 19. PMID 23182070
- [Background] Han SN, Gziri MM, Van Calsteren K, Amant F. Is chemotherapy during the first trimester of pregnancy really safe? Int J Cancer. 2013 Apr 1;132(7):1728. doi: 10.1002/ijc.27815. Epub 2012 Sep 28. No abstract available. PMID 22945483
- [Background] Han SN, Lotgerink A, Gziri MM, Van Calsteren K, Hanssens M, Amant F. Physiologic variations of serum tumor markers in gynecological malignancies during pregnancy: a systematic review. BMC Med. 2012 Aug 8;10:86. doi: 10.1186/1741-7015-10-86. PMID 22873292
- [Background] Loibl S, Han SN, Amant F. Being Pregnant and Diagnosed with Breast Cancer. Breast Care (Basel). 2012 Jun;7(3):204-209. doi: 10.1159/000339674. Epub 2012 Jun 27. PMID 22872793
- [Background] Amant F. Safety of chemotherapy in pregnancy. Clin Adv Hematol Oncol. 2012 Apr;10(4):258-9. No abstract available. PMID 22706488
- [Background] Verheecke M, Hermans E, Tuyaerts S, Souche E, Van Bree R, Verbist G, Everaert T, Cortes-Calabuig A, Van Houdt J, Van Calsteren K, Amant F. Acute Drug Effects on the Human Placental Tissue: The Development of a Placental Murine Xenograft Model. Reprod Sci. 2018 Dec;25(12):1637-1648. doi: 10.1177/1933719118756771. Epub 2018 Feb 13. PMID 29439620
- [Background] Boere I, Lok C, Vandenbroucke T, Amant F. Cancer in pregnancy: safety and efficacy of systemic therapies. Curr Opin Oncol. 2017 Sep;29(5):328-334. doi: 10.1097/CCO.0000000000000386. PMID 28614135
- [Background] Fruscio R, de Haan J, Van Calsteren K, Verheecke M, Mhallem M, Amant F. Ovarian cancer in pregnancy. Best Pract Res Clin Obstet Gynaecol. 2017 May;41:108-117. doi: 10.1016/j.bpobgyn.2016.09.013. Epub 2016 Oct 1. PMID 28029502
- [Background] Vercruysse DC, Deprez S, Sunaert S, Van Calsteren K, Amant F. Effects of prenatal exposure to cancer treatment on neurocognitive development, a review. Neurotoxicology. 2016 May;54:11-21. doi: 10.1016/j.neuro.2016.02.013. Epub 2016 Mar 4. PMID 26952827
- [Background] de Haan J, Vandecaveye V, Han SN, Van de Vijver KK, Amant F. Difficulties with diagnosis of malignancies in pregnancy. Best Pract Res Clin Obstet Gynaecol. 2016 May;33:19-32. doi: 10.1016/j.bpobgyn.2015.10.005. Epub 2015 Oct 19. PMID 26586541
- [Background] Han SN, Mhallem Gziri M, Van Calsteren K, Amant F. Cervical cancer in pregnant women: treat, wait or interrupt? Assessment of current clinical guidelines, innovations and controversies. Ther Adv Med Oncol. 2013 Jul;5(4):211-9. doi: 10.1177/1758834013494988. PMID 23858330
- [Background] Amant F, Han SN, Gziri MM, Dekrem J, Van Calsteren K. Chemotherapy during pregnancy. Curr Opin Oncol. 2012 Sep;24(5):580-6. doi: 10.1097/CCO.0b013e328354e754. PMID 22581358
- [Background] Amant F, Loibl S, Neven P, Van Calsteren K. Breast cancer in pregnancy. Lancet. 2012 Feb 11;379(9815):570-9. doi: 10.1016/S0140-6736(11)61092-1. PMID 22325662
- [Background] Han SN, Van Calsteren K, Amant F. Use of chemotherapy during pregnancy in the treatment of ovarian malignancies. Eur J Obstet Gynecol Reprod Biol. 2011 Jun;156(2):237. doi: 10.1016/j.ejogrb.2011.02.004. Epub 2011 Mar 25. No abstract available. PMID 21439708
- [Background] Amant F, Deckers S, Van Calsteren K, Loibl S, Halaska M, Brepoels L, Beijnen J, Cardoso F, Gentilini O, Lagae L, Mir O, Neven P, Ottevanger N, Pans S, Peccatori F, Rouzier R, Senn HJ, Struikmans H, Christiaens MR, Cameron D, Du Bois A. Breast cancer in pregnancy: recommendations of an international consensus meeting. Eur J Cancer. 2010 Dec;46(18):3158-68. doi: 10.1016/j.ejca.2010.09.010. PMID 20932740
- [Background] Amant F, Brepoels L, Halaska MJ, Gziri MM, Calsteren KV. Gynaecologic cancer complicating pregnancy: an overview. Best Pract Res Clin Obstet Gynaecol. 2010 Feb;24(1):61-79. doi: 10.1016/j.bpobgyn.2009.08.001. Epub 2009 Sep 8. PMID 19740709
- [Background] Van Calsteren K, Hartmann D, Van Aerschot L, Verbesselt R, Van Bree R, D'Hooge R, Amant F. Vinblastine and doxorubicin administration to pregnant mice affects brain development and behaviour in the offspring. Neurotoxicology. 2009 Jul;30(4):647-57. doi: 10.1016/j.neuro.2009.04.009. Epub 2009 May 5. PMID 19422850
- [Background] Amant F, Van Calsteren K, Halaska MJ, Beijnen J, Lagae L, Hanssens M, Heyns L, Lannoo L, Ottevanger NP, Vanden Bogaert W, Ungar L, Vergote I, du Bois A. Gynecologic cancers in pregnancy: guidelines of an international consensus meeting. Int J Gynecol Cancer. 2009 May;19 Suppl 1:S1-12. doi: 10.1111/IGC.0b013e3181a1d0ec. PMID 19509538
- [Background] Van Calsteren K, Devlieger R, De Catte L, D'Hooghe T, Chai DC, Mwenda JM, Vergote I, Amant F. Feasibility of ultrasound-guided percutaneous samplings in the pregnant baboon: a model for studies on transplacental transport. Reprod Sci. 2009 Mar;16(3):280-5. doi: 10.1177/1933719108324890. Epub 2008 Dec 15. PMID 19087981
- [Background] Amant F, Van Calsteren K, Vergote I, Ottevanger N. Gynecologic oncology in pregnancy. Crit Rev Oncol Hematol. 2008 Sep;67(3):187-95. doi: 10.1016/j.critrevonc.2008.01.006. Epub 2008 Mar 4. PMID 18296060
- [Result] Van Calsteren K, Heyns L, De Smet F, Van Eycken L, Gziri MM, Van Gemert W, Halaska M, Vergote I, Ottevanger N, Amant F. Cancer during pregnancy: an analysis of 215 patients emphasizing the obstetrical and the neonatal outcomes. J Clin Oncol. 2010 Feb 1;28(4):683-9. doi: 10.1200/JCO.2009.23.2801. Epub 2009 Oct 19. PMID 19841323
- [Result] Amant F, Van Calsteren K, Halaska MJ, Gziri MM, Hui W, Lagae L, Willemsen MA, Kapusta L, Van Calster B, Wouters H, Heyns L, Han SN, Tomek V, Mertens L, Ottevanger PB. Long-term cognitive and cardiac outcomes after prenatal exposure to chemotherapy in children aged 18 months or older: an observational study. Lancet Oncol. 2012 Mar;13(3):256-64. doi: 10.1016/S1470-2045(11)70363-1. Epub 2012 Feb 10. PMID 22326925
- [Result] Gziri MM, Debieve F, DE Catte L, Mertens L, Barrea C, VAN Calsteren K, Han SN, Heyns L, Amant F. Chemotherapy during pregnancy: effect of anthracyclines on fetal and maternal cardiac function. Acta Obstet Gynecol Scand. 2012 Dec;91(12):1465-8. doi: 10.1111/j.1600-0412.2012.01524.x. Epub 2012 Nov 1. PMID 22880883
- [Result] Loibl S, Han SN, von Minckwitz G, Bontenbal M, Ring A, Giermek J, Fehm T, Van Calsteren K, Linn SC, Schlehe B, Gziri MM, Westenend PJ, Muller V, Heyns L, Rack B, Van Calster B, Harbeck N, Lenhard M, Halaska MJ, Kaufmann M, Nekljudova V, Amant F. Treatment of breast cancer during pregnancy: an observational study. Lancet Oncol. 2012 Sep;13(9):887-96. doi: 10.1016/S1470-2045(12)70261-9. Epub 2012 Aug 16. PMID 22902483
- [Result] Gziri MM, Amant F, Debieve F, Van Calsteren K, De Catte L, Mertens L. Effects of chemotherapy during pregnancy on the maternal and fetal heart. Prenat Diagn. 2012 Jul;32(7):614-9. doi: 10.1002/pd.3847. Epub 2012 Apr 17. PMID 22508540
- [Result] Mhallem Gziri M, Han SN, Van Calsteren K, Heyns L, Delaere P, Nuyts S, Van den Heuvel F, Cheron AC, Fossion E, Van den Weyngaert D, Lok C, Amant F. Tongue cancers during pregnancy: Case reports and review of literature. Head Neck. 2013 Apr;35(4):E102-8. doi: 10.1002/hed.21924. Epub 2011 Oct 19. PMID 22009853
- [Result] Gziri MM, Hui W, Amant F, Van Calsteren K, Ottevanger N, Kapusta L, Mertens L. Myocardial function in children after fetal chemotherapy exposure. A tissue Doppler and myocardial deformation imaging study. Eur J Pediatr. 2013 Feb;172(2):163-70. doi: 10.1007/s00431-012-1849-7. Epub 2012 Oct 5. PMID 23052619
- [Result] Boussios S, Han SN, Fruscio R, Halaska MJ, Ottevanger PB, Peccatori FA, Koubkova L, Pavlidis N, Amant F. Lung cancer in pregnancy: report of nine cases from an international collaborative study. Lung Cancer. 2013 Dec;82(3):499-505. doi: 10.1016/j.lungcan.2013.09.002. Epub 2013 Sep 12. PMID 24091171
- [Result] Amant F, von Minckwitz G, Han SN, Bontenbal M, Ring AE, Giermek J, Wildiers H, Fehm T, Linn SC, Schlehe B, Neven P, Westenend PJ, Muller V, Van Calsteren K, Rack B, Nekljudova V, Harbeck N, Untch M, Witteveen PO, Schwedler K, Thomssen C, Van Calster B, Loibl S. Prognosis of women with primary breast cancer diagnosed during pregnancy: results from an international collaborative study. J Clin Oncol. 2013 Jul 10;31(20):2532-9. doi: 10.1200/JCO.2012.45.6335. Epub 2013 Apr 22. PMID 23610117
- [Result] Verheecke M, Halaska MJ, Lok CA, Ottevanger PB, Fruscio R, Dahl-Steffensen K, Kolawa W, Gziri MM, Han SN, Van Calsteren K, Van den Heuvel F, De Vleeschouwer S, Clement PM, Menten J, Amant F; ESGO Task Force 'Cancer in Pregnancy'. Primary brain tumours, meningiomas and brain metastases in pregnancy: report on 27 cases and review of literature. Eur J Cancer. 2014 May;50(8):1462-71. doi: 10.1016/j.ejca.2014.02.018. Epub 2014 Mar 14. PMID 24636876
- [Result] Vandenbroucke T, Van Calsteren K, Amant F. Pediatric Outcome after Maternal Cancer Diagnosed during Pregnancy. N Engl J Med. 2016 Feb 18;374(7):693. doi: 10.1056/NEJMc1515462. No abstract available. PMID 26886537
- [Result] Amant F, Vandenbroucke T, Verheecke M, Fumagalli M, Halaska MJ, Boere I, Han S, Gziri MM, Peccatori F, Rob L, Lok C, Witteveen P, Voigt JU, Naulaers G, Vallaeys L, Van den Heuvel F, Lagae L, Mertens L, Claes L, Van Calsteren K; International Network on Cancer, Infertility, and Pregnancy (INCIP). Pediatric Outcome after Maternal Cancer Diagnosed during Pregnancy. N Engl J Med. 2015 Nov 5;373(19):1824-34. doi: 10.1056/NEJMoa1508913. Epub 2015 Sep 28. PMID 26415085
- [Result] Loibl S, Schmidt A, Gentilini O, Kaufman B, Kuhl C, Denkert C, von Minckwitz G, Parokonnaya A, Stensheim H, Thomssen C, van Calsteren K, Poortmans P, Berveiller P, Markert UR, Amant F. Breast Cancer Diagnosed During Pregnancy: Adapting Recent Advances in Breast Cancer Care for Pregnant Patients. JAMA Oncol. 2015 Nov;1(8):1145-53. doi: 10.1001/jamaoncol.2015.2413. PMID 26247818
- [Result] Vandenbroucke T, Amant F. Development of children born to mothers with cancer during pregnancy: comparing in utero chemotherapy-exposed children with nonexposed controls. Am J Obstet Gynecol. 2015 Jun;212(6):830-1. doi: 10.1016/j.ajog.2015.01.035. Epub 2015 Jan 28. No abstract available. PMID 25637847
- [Result] Vandenbroucke T, Verheecke M, Van Calsteren K, Han S, Claes L, Amant F. Fetal outcome after prenatal exposure to chemotherapy and mechanisms of teratogenicity compared to alcohol and smoking. Expert Opin Drug Saf. 2014 Dec;13(12):1653-65. doi: 10.1517/14740338.2014.965677. Epub 2014 Nov 10. PMID 25382454
- [Result] van Hasselt JGC, van Calsteren K, Heyns L, Han S, Mhallem Gziri M, Schellens JHM, Beijnen JH, Huitema ADR, Amant F. Optimizing anticancer drug treatment in pregnant cancer patients: pharmacokinetic analysis of gestation-induced changes for doxorubicin, epirubicin, docetaxel and paclitaxel. Ann Oncol. 2014 Oct;25(10):2059-2065. doi: 10.1093/annonc/mdu140. Epub 2014 Apr 8. PMID 24713311
- [Result] Dekrem J, Van Calsteren K, Amant F. Effects of fetal exposure to maternal chemotherapy. Paediatr Drugs. 2013 Oct;15(5):329-34. doi: 10.1007/s40272-013-0040-6. PMID 23856754
- [Result] Gziri MM, Pokreisz P, De Vos R, Verbeken E, Debieve F, Mertens L, Janssens SP, Amant F. Fetal rat hearts do not display acute cardiotoxicity in response to maternal Doxorubicin treatment. J Pharmacol Exp Ther. 2013 Sep;346(3):362-9. doi: 10.1124/jpet.113.205419. Epub 2013 Jun 21. PMID 23792410
- [Result] de Haan J, Verheecke M, Van Calsteren K, Van Calster B, Shmakov RG, Mhallem Gziri M, Halaska MJ, Fruscio R, Lok CAR, Boere IA, Zola P, Ottevanger PB, de Groot CJM, Peccatori FA, Dahl Steffensen K, Cardonick EH, Polushkina E, Rob L, Ceppi L, Sukhikh GT, Han SN, Amant F; International Network on Cancer and Infertility Pregnancy (INCIP). Oncological management and obstetric and neonatal outcomes for women diagnosed with cancer during pregnancy: a 20-year international cohort study of 1170 patients. Lancet Oncol. 2018 Mar;19(3):337-346. doi: 10.1016/S1470-2045(18)30059-7. Epub 2018 Jan 26. PMID 29395867
- [Result] de Haan J, van Thienen JV, Casaer M, Hannivoort RA, Van Calsteren K, van Tuyl M, van Gerwen MM, Debeer A, Amant F, Painter RC. Severe Adverse Reaction to Vemurafenib in a Pregnant Woman with Metastatic Melanoma. Case Rep Oncol. 2018 Feb 15;11(1):119-124. doi: 10.1159/000487128. eCollection 2018 Jan-Apr. PMID 29606950
- [Result] Boucek J, de Haan J, Halaska MJ, Plzak J, Van Calsteren K, de Groot CJM, Dahl Steffensen K, Fruscio R, Massolt ET, Klaritsch P, Zola P, Amant F; International Network on Cancer, Infertility, and Pregnancy. Maternal and obstetrical outcome in 35 cases of well-differentiated thyroid carcinoma during pregnancy. Laryngoscope. 2018 Jun;128(6):1493-1500. doi: 10.1002/lary.26936. Epub 2017 Oct 8. PMID 28988434
- [Result] de Haan J, Lok CA, de Groot CJ, Crijns MB, Van Calsteren K, Dahl Steffensen K, Halaska MJ, Altintas S, Boere IA, Fruscio R, Kolawa W, Witteveen PO, Amant F; International Network on Cancer, Infertility and Pregnancy (INCIP). Melanoma during pregnancy: a report of 60 pregnancies complicated by melanoma. Melanoma Res. 2017 Jun;27(3):218-223. doi: 10.1097/CMR.0000000000000327. PMID 28099365
- [Result] Verheecke M, Cortes Calabuig A, Finalet Ferreiro J, Brys V, Van Bree R, Verbist G, Everaert T, Leemans L, Gziri MM, Boere I, Halaska MJ, Vanhoudt J, Amant F, Van Calsteren K. Genetic and microscopic assessment of the human chemotherapy-exposed placenta reveals possible pathways contributive to fetal growth restriction. Placenta. 2018 Apr;64:61-70. doi: 10.1016/j.placenta.2018.03.002. Epub 2018 Mar 9. PMID 29626982
- [Result] Vandenbroucke T, Verheecke M, Fumagalli M, Lok C, Amant F. Effects of cancer treatment during pregnancy on fetal and child development. Lancet Child Adolesc Health. 2017 Dec;1(4):302-310. doi: 10.1016/S2352-4642(17)30091-3. Epub 2017 Sep 29. PMID 30169185
- [Result] Gziri MM, Brunee L, Cayphas C, Prigogine T, Van Raemdonck D, Amant F, Hubinont C. Low-grade bronchial mucoepidermoid carcinoma during pregnancy successfully treated by lobectomy. J Obstet Gynaecol. 2017 Nov;37(8):1082-1084. doi: 10.1080/01443615.2017.1308325. Epub 2017 Jun 1. No abstract available. PMID 28569562
- [Result] de Haan J, Van Calsteren K, Lok CAR, de Groot CJM, Amant F. Comment on "Maternal and perinatal outcomes in pregnancy-associated melanoma. Report of two cases and a systematic literature review". Eur J Obstet Gynecol Reprod Biol. 2017 Sep;216:261-262. doi: 10.1016/j.ejogrb.2017.07.025. Epub 2017 Jul 23. No abstract available. PMID 28768572
- [Result] Vandenbroucke T, Han SN, Van Calsteren K, Wilderjans TF, Van den Bergh BRH, Claes L, Amant F. Psychological distress and cognitive coping in pregnant women diagnosed with cancer and their partners. Psychooncology. 2017 Aug;26(8):1215-1221. doi: 10.1002/pon.4301. Epub 2016 Nov 21. PMID 27859911
- [Result] Gziri MM, Han SN, Amant F. Use of general anesthesia and sentinel node procedure during pregnancy. J Surg Oncol. 2012 Dec;106(8):1008. doi: 10.1002/jso.23164. Epub 2012 Jun 4. No abstract available. PMID 22674350
- [Result] Lambrechts S, Van Calsteren K, Capoen A, Op De Beeck K, Joniau S, Timmerman D, Amant F. Polypoid endometriosis of the bladder during pregnancy mimicking urachal carcinoma. Ultrasound Obstet Gynecol. 2011 Oct;38(4):475-8. doi: 10.1002/uog.8985. Epub 2011 Sep 6. PMID 21374752
- [Result] Van Calsteren K, Verbesselt R, Van Bree R, Heyns L, de Bruijn E, de Hoon J, Amant F. Substantial variation in transplacental transfer of chemotherapeutic agents in a mouse model. Reprod Sci. 2011 Jan;18(1):57-63. doi: 10.1177/1933719110379650. Epub 2010 Sep 8. PMID 20826505
- [Result] Van Calsteren K, Verbesselt R, Beijnen J, Devlieger R, De Catte L, Chai DC, Van Bree R, Heyns L, de Hoon J, Amant F. Transplacental transfer of anthracyclines, vinblastine, and 4-hydroxy-cyclophosphamide in a baboon model. Gynecol Oncol. 2010 Dec;119(3):594-600. doi: 10.1016/j.ygyno.2010.08.019. Epub 2010 Sep 17. PMID 20846713
- [Result] Calsteren KV, Verbesselt R, Devlieger R, De Catte L, Chai DC, Van Bree R, Heyns L, Beijnen J, Demarsin S, de Bruijn E, de Hoon J, Amant F. Transplacental transfer of paclitaxel, docetaxel, carboplatin, and trastuzumab in a baboon model. Int J Gynecol Cancer. 2010 Dec;20(9):1456-64. doi: 10.1111/IGC.0b013e3181fb18c8. PMID 21307819
- [Result] Van Calsteren K, Verbesselt R, Ottevanger N, Halaska M, Heyns L, Van Bree R, de Bruijn E, Chai D, Delforge M, Noens L, Renard V, Witteveen E, Rob L, de Hoon J, Amant F. Pharmacokinetics of chemotherapeutic agents in pregnancy: a preclinical and clinical study. Acta Obstet Gynecol Scand. 2010 Oct;89(10):1338-45. doi: 10.3109/00016349.2010.512070. PMID 20846067
- [Result] Van Calsteren K, Hanssens M, Moerman P, Orye G, Bielen D, Vergote I, Amant F. Successful conservative treatment of endocervical adenocarcinoma stage Ib1 diagnosed early in pregnancy. Acta Obstet Gynecol Scand. 2008;87(2):250-3. doi: 10.1080/00016340701870794. PMID 18231896
- [Result] Van Calsteren K, Van Mensel K, Joniau S, Oyen R, Hanssens M, Amant F, Van Poppel H. Urachal carcinoma during pregnancy. Urology. 2006 Jun;67(6):1290.e19-21. doi: 10.1016/j.urology.2005.12.041. PMID 16750250
- [Derived] Kruse AM, Huis In 't Veld EA, van Grotel M, Amant F, van Tinteren H, van den Heuvel-Eibrink MM, Verwaaijen EJ. Motor development in toddlers prenatally exposed to maternal cancer treatment: a national cohort study in the Netherlands. EClinicalMedicine. 2026 Jan 17;92:103738. doi: 10.1016/j.eclinm.2025.103738. eCollection 2026 Feb. PMID 41623857
- [Derived] Van Assche IA, Van Calsteren K, Huis In 't Veld EA, van Gerwen M, Heylen L, LeJeune CL, Cardonick E, Halaska MJ, Fruscio R, Fumagalli M, van Dijk-Lokkart EM, Lemiere J, van Grotel M, Lagae L, van den Heuvel-Eibrink MM, Amant F. Child outcomes after prenatal exposure to platinum and taxane-based chemotherapy: an unplanned interim analysis of the international network on cancer, infertility, and pregnancy study. EClinicalMedicine. 2024 Nov 11;78:102922. doi: 10.1016/j.eclinm.2024.102922. eCollection 2024 Dec. PMID 39588212
- [Derived] Vandenbroucke T, Verheecke M, van Gerwen M, Van Calsteren K, Halaska MJ, Fumagalli M, Fruscio R, Gandhi A, Veening M, Lagae L, Ottevanger PB, Voigt JU, de Haan J, Gziri MM, Maggen C, Mertens L, Naulaers G, Claes L, Amant F; International Network on Cancer, Infertility and Pregnancy (INCIP). Child development at 6 years after maternal cancer diagnosis and treatment during pregnancy. Eur J Cancer. 2020 Oct;138:57-67. doi: 10.1016/j.ejca.2020.07.004. Epub 2020 Aug 25. PMID 32858478
- See also: This site provides background information on the problem of cancer in pregnancy and details further the project. — http://www.cancerinpregnancy.org